CLINICAL TRIAL: NCT07141550
Title: The Effect of Kinesthetic Brain Exercises Applied in Addition to Telerehabilitation-Based Pilates Exercises on Cognitive Functions, Symptom Management, Functional Performance, and Quality of Life in Women With Fibromyalgia
Brief Title: Kinesthetic Brain and Telerehab Pilates for Cognitive and Functional Outcomes in Women With Fibromyalgia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Democracy University (Other)
Responsible Party: Principal Investigator, Betül Taşpınar, Prof. Dr., Izmir Democracy University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Fibromyalgia
Record Dates: First submitted 2025-08-19; First posted 2025-08-26 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Fibromyalgia
Keywords: fibromyalgia; telerehabilitation; pilates-based exercises; kinesthetic brain exercises
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- İntervention group (Other): Clinical pilates and kinesthetic brain exercises will be applied to this group
  Interventions: Other: Clinical Pilates Group; Other: Kinesthetic Brain Exercises Group
- Control Group (Other): group to receive clinical Pilates
  Interventions: Other: Clinical Pilates Group

INTERVENTIONS:
Other: Clinical Pilates Group — Participants will be introduced to the principles of Pilates, the workout program, and its five key elements: neutral spine, lumbopelvic and scapular stabilization, focus, and breathing. Clinical Pilates sessions will be held twice weekly for 8 weeks, 60 minutes each, via synchronous telerehabilitation (Zoom/WhatsApp). Each session includes a 10-minute warm-up, 40 minutes of Pilates exercises, and a 10-minute cool-down. The physiotherapist will provide visual and verbal guidance to ensure correct posture and breathing. Exercises start with 6-8 repetitions in the first week, increasing progressively according to participant ability and advancing to higher-level positions.
  Other Names: CGP
Other: Kinesthetic Brain Exercises Group — 16 sessions, approximately 40 minutes each, will be administered twice a week for eight weeks by a physical therapist via video chat programs such as Zoom or WhatsApp. Kinesthetic brain exercises consist of three phases: a warm-up phase, an exercise phase, and a cool-down phase. The warm-up and cool-down phases consist of hand-eye coordination and relaxation exercises. The exercise phase consists of independent and dependent movements, as well as a combination of both.
  Other Names: KBE
  Arms: İntervention group

SUMMARY:
Fibromyalgia is a chronic pain syndrome often accompanied by fatigue, psychological problems, and cognitive dysfunction, leading to reduced quality of life. Telerehabilitation-based Pilates has been shown to improve symptoms and function in fibromyalgia, while kinesthetic brain exercises may enhance cognitive performance through neuroplasticity. This study aims to evaluate the effects of adding kinesthetic brain exercises to telerehabilitation-based Pilates on cognitive functions, symptom management, functional performance, and quality of life in women with fibromyalgia.

DETAILED DESCRIPTION:
Fibromyalgia (FM) is a chronic and widespread pain syndrome affecting the musculoskeletal system. It is the second most common rheumatic disease worldwide and is associated with pain, fatigue, sleep disturbance, morning stiffness, psychological problems, and cognitive dysfunction. These symptoms contribute to physical disability, reduced physical activity, and difficulties in social and occupational life. The pathophysiology of FM is not clearly defined, but central sensitization is thought to play a key role. The unclear etiology and the limited effectiveness of existing treatment methods make the management of FM challenging and highlight the need for multidisciplinary treatment approaches.

Cognitive impairment, commonly referred to as "fibro-fog," is observed in more than half of individuals with FM. It negatively affects attention, perception, and executive functions, thereby reducing daily functioning and overall quality of life. For this reason, therapeutic strategies targeting cognitive functions in FM have gained increasing importance. Neuroplasticity, the brain's ability to adapt to environmental changes and experiences, is a promising mechanism for improving cognitive functions. Regular exercise has been shown to stimulate neuroplasticity and enhance cognition.

In recent years, telerehabilitation has become a valuable treatment option, especially for individuals with chronic diseases who cannot access regular healthcare services. It provides an effective, safe, and accessible method for assessment, intervention, education, and monitoring, while also saving time and cost. Telerehabilitation has been demonstrated to improve pain, functional capacity, quality of life, and treatment adherence in patients with FM.

Exercise therapy remains a cornerstone in FM management. Pilates, as a mind-body exercise focusing on controlled movement, stretching, and breathing, aims to strengthen core muscles, improve posture, flexibility, and balance, and enhance overall physical and psychological well-being. It can be adapted to individual needs, making it a suitable component of multidisciplinary treatment programs. Clinical studies indicate that Pilates is effective in reducing pain, improving muscle strength, posture, and function, and enhancing quality of life in FM.

Kinesthetic brain exercises, which combine movement and mental tasks, are designed to target cognitive processes such as attention, memory, and problem solving. By supporting motor learning and neuroplasticity, they may improve synaptic reorganization and enhance cognitive as well as physical performance. Given that FM affects both mental and physical functioning, kinesthetic brain exercises may represent a promising complementary approach.

To date, no studies have investigated the combined effects of kinesthetic brain exercises and telerehabilitation-based Pilates in women with fibromyalgia. This study aims to evaluate the effectiveness of adding kinesthetic brain exercises to a telerehabilitation-based Pilates program on cognitive functions, symptom management, functional performance, and quality of life in women with FM.

ELIGIBILITY:
Inclusion Criteria:

* • Individuals aged 18-65

  * Volunteering
  * Female
  * Individuals diagnosed with fibromyalgia according to the 2016 American College of Rheumatology (ACR) criteria
  * Possessing the necessary infrastructure (internet) and equipment (smartphone, tablet, or computer) for telerehabilitation

Exclusion Criteria:

* • Having a severe reading comprehension problem

  * Having a severe vision or hearing problem
  * Being pregnant
  * Having an active infection
  * Having a neurological or orthopedic problem that prevents mobility
  * Having any rheumatic disease other than fibromyalgia
  * Having cancer
  * Having undergone major surgery within the last 6 months
  * Individuals with psychiatric or cognitive disorders that would prevent measurements from being taken in the study

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-03-25 (Estimated); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment Scale | At baseline and after 8 weeks
  This is a sensitive assessment scale used to assess cognitive functions. It assesses visual-spatial perception, executive functions, naming, memory, attention, language, abstract thinking, delayed recall, and orientation functions (Selekler et al., 2010). The scale consists of 11 items, and the maximum score is 30. A score of 21 or less indicates cognitive dysfunction.
Stroop Test | At baseline and after 8 weeks
  The Stroop Test reflects frontal region activity and is considered the gold standard for measuring attention. A study by Karakaş et al. determined its reliability and validity in Turkish culture. The Stroop test consists of four sheets of paper measuring 14.0 cm x 21.5 cm. Each sheet contains a total of 24 randomly written words in 6 rows and 4 columns. The test consists of five parts, and each part is scored separately. The first sheet requires reading words written in black; the second sheet requires reading words written in color; the third sheet requires saying the colors of circular shapes; the fourth sheet requires saying only the color of unrelated words written in color without reading them; and the fifth sheet requires correctly saying the color of words printed in a color different from the original. Scoring is based on time, the number of errors, and corrected errors
Trail Making Test | at baseline and after 8 weeks.
  The Trail Making Test (TMT) is a two-part test used to assess executive functions, measuring visual-motor skills, processing speed, attention, planning, and set-shifting abilities. In Part A, participants are asked to connect sequential numbers from 1 to 25 in circles, while Part B asks participants to match numbers and letters sequentially (1-A-2-B). Part A assesses processing speed, while Part B assesses set-shifting and sequential thinking skills. Completion times for both sections are recorded
Forward-backward digit span test | at baseline and after 8 weeks.
  It is a short and easy-to-administer test that assesses short-term memory and attention. It consists of two parts: a forward digit span test and a backward digit span test. The forward counting test begins with two 3-digit items and ends with two 9-digit items. The backward counting test begins with two 2-digit items and ends with two 8-digit items. Two attempts are allowed. The maximum score for forward digit span is 8, and for backward digit span, it is 7, for a total of 15 points. Generally, the difference between the forward and backward digit span results is expected to be two
Visual Analog Scale (VAS) | at baseline and after 8 weeks.
  It is frequently preferred because it is an easy and understandable scale. Participants are asked to mark the appropriate location for their pain intensity on a 10-cm horizontal line, with the beginning representing no pain and the end representing unbearable pain. Pain ranges are as follows: <3 indicates mild pain, 3-6 indicates moderate pain, and >6 indicates severe pain. Pain will also be assessed in four different situations: night pain, daytime pain, pain at rest, and activity pain.
The Pain Catastrophizing Scale | at baseline and after 8 weeks.
  The Pain Catastrophizing Scale is a self-administered questionnaire used to assess patients' thoughts and feelings about pain. Developed by Sullivan and colleagues in 1995, it is a reliable and valid questionnaire for Turkish that assesses specific variables such as severe pain, disability, and emotional disturbance following trauma or tissue damage. It consists of subscales for "helplessness" (inability to cope effectively with pain), "magnification" (displeasure caused by excessive focus on the negative consequences of pain), and "rumination" (inability to inhibit pain-related thoughts). It consists of 13 items and is scored from 0 to 4. It has a total of 52 points
Evaluation of fatigue | at baseline and after 8 weeks.
  Fatigue severity will be assessed using the Visual Analog Scale (VAS). It is frequently preferred because it is an easy and understandable scale. The beginning indicates no fatigue, and the end indicates extreme fatigue. To measure severity, a ruler will be used to measure the severity from the beginning of the line to the point marked by the participant and recorded
Multidimensional Fatigue Inventory-20 (MFI-20) | at baseline and after 8 weeks.
  General fatigue, physical fatigue, mental fatigue, decreased motivation, and decreased activity. It has been used in various descriptive and experimental studies of many different diseases, including fibromyalgia. When completing the scale, participants are asked to select the rating closest to their level, from "no" to "yes" to "very true" out of 5. It consists of 20 questions. A high score indicates severe fatigue
Assessment of disease severity | at baseline and after 8 weeks.
  It is a self-reported questionnaire that measures functional capacity and disease severity in patients with fibromyalgia. It is an easy and short-term questionnaire. It consists of 21 questions in three sections covering function, global impact, and symptoms. It concerns experiences over the past 7 days and is scored using an 11-point numerical rating scale. It consists of a total score for the function domain (range 0 to 90, divided by 3), a global impact score (range 0 to 20), and a symptoms domain score (range 0 to 100, divided by 2)
Timed Up and Go Test | at baseline and after 8 weeks.
  It is a reliable test frequently used to assess agility, dynamic balance, and functional mobility in individuals with fibromyalgia This test begins with the patient sitting in a chair with a backrest. The patient stands up from the chair, walks to a marker 3 meters away, and records the time they return to their seat. It will be administered three times, and the best value will be recorded
Trunk flexor endurance test | at baseline and after 8 weeks.
  The participant will be positioned with their back supported, with their knees at 90 degrees and their torso at 60 degrees, their back straight, and their hands crossed on opposite shoulders. The physiotherapist will stabilize the feet and ask the participant to maintain this position as much as possible, removing the back support. The test will be terminated when the trunk angle is observed to disappear, and the elapsed time in seconds will be recorded.
Trunk extensor endurance test | at baseline and after 8 weeks.
  The test begins when the subject, lying face down on a stretcher, with ankles and knees fixed on the stretcher, the trunk hanging from the stretcher with the spina iliaca anterior superior (SIAS) positioned over the edge of the stretcher, and the hands crossed in front of the stretcher, holding the shoulders, reaches a horizontal position. The time the subject maintains this position is recorded in seconds
Lateral Trunk Endurance Test | at baseline and after 8 weeks.
  The test will begin in a side-lying position. The participant will be asked to position their knees straight, their feet in a tandem stance, with the front foot on top, supporting their body with their bottom elbow and placing their top elbow on the opposite shoulder. They will be instructed to use only three points of support (elbows and feet) when lifting their hips off the mat. The test will end when the hips approach the mat or when support is gained from another location, and the elapsed time will be recorded
Plank | At baseline and after 8 weeks
  To evaluate the plank test, the time spent in push-up position on the floor mat, with the toes fixed on the floor mat, elbows flexed, touching the floor mat and hips up, without changing the position, will be recorded in seconds
Assessment of Biopsychosocial Status | At baseline and after 8 weeks
  The Cognitive Exercise Therapy Approach-Biopsychosocial Scale, which Zahid and Ünal developed in 2018 and has proven valid and reliable in individuals with fibromyalgia, will be used. This 30-item scale assesses the biopsychosocial processes associated with the disease. A 5-point Likert-type score is used for scoring the scale. A total score is obtained by scoring items as follows: No never = 0, Yes rarely = 1, Yes sometimes = 2, Yes often = 3, and Yes always = 4. A higher score indicates a lower biopsychosocial status
Quality of Life Assessment | at baseline and after 8 weeks.
  The Short Form-36 Quality of Life scale, consisting of 36 questions and will be used to assess participants' quality of life. This questionnaire examines eight dimensions of health with 36 items: social function, physical function, physical role difficulty, energy, mental health, emotional role difficulty, general health perception, and pain. In the absence of any limitations or barriers, the maximum possible score is 100. Each dimension is assessed independently, with a higher score indicating a higher quality of life for that dimension

CONTACTS AND LOCATIONS:
Overall Officials: Onur Engin, Assist.Prof, Principal Investigator — Izmir Democracy University; Ferruh Taspinar, Prof.Dr., Principal Investigator — Izmir Democracy University